CLINICAL TRIAL: NCT02794155
Title: Phase 2b, Multicenter, Randomized, Double Blind, Titration Trial for Efficacy and Safety of HDV Insulin Lispro in Combination With a Basal Insulin Versus Insulin Lispro in Combination With a Basal Insulin in Patients With Type 1 Diabetes
Brief Title: Study of HDV Insulin Versus Insulin in Type 1 Diabetes Subjects (ISLE-1)
Acronym: ISLE-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Diasome Pharmaceuticals (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DP 01-2015-01
Record Dates: First submitted 2016-05-16; First posted 2016-06-08 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2017-01

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Group (Experimental): HDV Insulin Lispro subcutaneous, pre-prandial dosing, 26 week treatment period
  Interventions: Drug: HDV Insulin Lispro
- Control Group (Active Comparator): Insulin Lispro subcutaneous, Pre-prandial dosing, 26 week treatment period
  Interventions: Drug: Insulin LISPRO

INTERVENTIONS:
Drug: HDV Insulin Lispro — HDV Insulin Lispro: ~1% of the Insulin Lispro is bound to HDV (Hepatocyte Directed Vesicle)
  Other Names: HDV Humalog
  Arms: Test Group
Drug: Insulin LISPRO — Insulin Lispro: no bound insulin
  Other Names: Humalog
  Arms: Control Group

SUMMARY:
This will be a Phase 2b, multicenter, randomized, double blind, titration clinical study, evaluating the efficacy and safety in the HDV Insulin Lispro Group versus Insulin Lispro Group in patients with type 1 diabetes over a 26 week treatment period. The patients will be randomized using a centrally allocated randomization scheme to 1 of the 2 treatment arms in an overall 2:1 scheme (HDV Insulin Lispro: Insulin Lispro). Both arms will receive the randomized treatment in combination with glargine or detemir. Goal to demonstrate that the efficacy of HDV insulin lispro administered in combination with a basal insulin (HDV Insulin Lispro group) is non-inferior to insulin lispro in combination with a basal insulin (Insulin Lispro group), in effects on glycated hemoglobin (HbA1c) in patients with type 1 diabetes. If non-inferiority is demonstrated, confirm that HDV insulin lispro in combination with a basal insulin (HDV Insulin Lispro group) is superior to insulin lispro in combination with a basal insulin (Insulin Lispro group), in effects on HbA1c in patients with type 1 diabetes (≥ 0.4% decrease in HbA1c).

DETAILED DESCRIPTION:
This will be a Phase 2b, multicenter, randomized, double blind, titration clinical study, evaluating the efficacy and safety in the HDV Insulin Lispro Group versus Insulin Lispro Group in patients with type 1 diabetes over a 26 week treatment period. The patients will be randomized using a centrally allocated randomization scheme to 1 of the 2 treatment arms in an overall 2:1 scheme (HDV Insulin Lispro: Insulin Lispro). Both arms will receive the randomized treatment in combination with glargine or detemir.

SCREENING (Visit 1, Week -4 to -1) Patients will arrive for Screening following an 8 hour fast. During Screening, patients will sign the informed consent form, be reviewed for inclusion/exclusion, and provide medical history, concomitant medications, and demographics. They will have a brief physical exam and provide vital signs. Safety hematology/chemistry/urinalysis (with liver enzymes) will include infectious serology, and serum pregnancy test for women of childbearing potential. An ECG will be performed and patients will provide samples for HbA1c determination.

Patients taking lispro/glargine or lispro/detemir at the time of Screening and who meet all eligibility criteria will proceed to Visit 2 (Week -1).

TREATMENT PERIOD Visit 1a (Week -2) will be required only if a patient must convert to lispro prior to Visit 3 (Week 0, randomization). Patients taking non-lispro/glargine or non-lispro/detemir or using an insulin pump will be converted to lispro/glargine or lispro/detemir (respectively) using equivalent insulin units, then proceed to Visit 2 (Week -1) after 1 week on the new regimen. At Visit 2 (Week -1), patients will receive the CGM and be trained on its use. Patients will also have their first Mixed Meal Tolerance Test (MMTT) during Visit 2 (Week -1) accompanied by monitoring of blood ketones pre- and post-ingestion. CGM and MMTT will be repeated at Visits 9 (Week 12) and 14 (Week 25). A diary, glucose meter, and supplies will also be provided at Visit 2 (Week -1). Patients will be instructed on how to perform self-monitored blood glucose measurements (SMBG). During Visit 3 (Week 0), eligible patients will be randomized by IWRS to either treatment arm (Test Group or Control Group) and baseline data will be collected. All visits will include progress reviews and safety procedures. Safety hematology/chemistry/ urinalysis at Visits 2 (Week -1), 10 (Week 13), 14 (Week 25) and 16 (Week 27) will include liver enzymes. At Visits 6 (Week 5) and 12 (Week 19), liver enzymes will be the only chemistry safety tests performed. The only chemistry safety tests performed at Visits 2 (Week -1), 9 (Week 12), and 14 (Week 25) will be blood ketones; these will be measured at baseline and 3 hours after the MMTT. HbA1c will be measured at Visits 3 (Week 0), 4 (Week 1), 7 (Week 7), 10 (Week 13), 12 (Week 19), and 15 (Week 26). Fasting blood glucose will be measured at Visits 3 (Week 0), 10 (Week 13), and 15 (Week 26). An in-clinic urine pregnancy test will be performed at all visits for women of childbearing potential. MRI will be performed at Visits 3 (Week 0) and 14 (Week 25) for approximately 20% of patients in each treatment arm. MRI may also be performed on a case-by-case basis in the event of abnormal liver enzyme results. Patients will receive weekly telephone calls from the PI or a designee to discuss insulin dosing and titration.

FOLLOW-UP Visit 16 (Week 27) is a safety follow-up visit which will include a physical exam. Safety hematology/chemistry/ urinalysis (including liver enzymes) will include a urine pregnancy test for women of childbearing potential.

Concomitant medications, vital signs, and adverse events will be recorded throughout the entire study period.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 yrs. of age
2. Clinical diagnosis of Type 1 diabetes mellitus for at least 12 months
3. Body Mass Index (BMI) ≤ 35 Kg/m2
4. Basal insulin includes insulin Glargine or insulin Detemir
5. Patient should be using bolus insulin defined as 2 to 4 doses of regular human insulin or rapid-acting analog at meals
6. HbA1c ≥ 7.0% and ≤ 10.5%
7. Fasting C-peptide ≤ 0.5 pmol/mL
8. Willingness to adhere to protocol and perform all required tests
9. Willing and able to review and sign the Informed Consent Form.
10. If child bearing age, must use acceptable form of birth control (ligation, 2 forms of birth control)
11. Willing to wear CGM devices and complete diaries.

Exclusion Criteria:

1. Total daily insulin dose ≥ 1.5 IU/kg/day.
2. History of recent blood transfusions (within previous 3 months), hemoglobinopathies, or any other conditions that effect HbA1c measurements
3. Evidence of serious complications of diabetes (eg, Symptomatic autonomic neuropathy)
4. Patients who are selected to but are unwilling or unable to participate in the MRI evaluation subset. (These patients may still participate in the non-MRI subset).
5. Significant cardiovascular dysfunction or history within 12 months of Screening, eg, congestive heart failure (New York Heart Association Class III or IV), or clinically significant arrhythmia, myocardial infarction, cardiac surgery; history of valvular heart disease including mild or greater aortic insufficiency, or moderate or greater mitral insufficiency; recurrent syncope, transient ischemic attacks, or cerebrovascular accident
6. Impaired liver function with elevated enzymes > 50% above the normal range at Screening. Patients with elevated liver enzymes may have the test repeated only at Visit 2 on a case-by-case basis at the request of the PI.
7. Creatinine level > 2 mg/dL for men, and > 1.8 mg/dL for women at Screening.
8. Patient on low carbohydrate diet, such as Atkins Diet
9. History of Adrenal supplementation within 3 years of Screening.
10. History of unawareness or SEVERE recurrent hypoglycemia, defined as a patient who is unaware of symptoms of hypoglycemia, or due to autonomic dysfunction, has no inherent warnings of hypoglycemia, and therefore requires outside assistance to rectify any episodes of hypoglycemia
11. Patients treated with systemic corticosteroids (Sporadic use of inhaled, intraarticular, and topical corticosteroids is not considered systemic).
12. Patients with triglyceride levels ≥500 mg/dL at Screening.
13. Patients with a history of cancer within the past 5 years, excluding basal or squamous cell carcinoma localized to the skin.
14. Epilepsy or other physical or medical conditions which could result in non-compliance with the study.
15. Participation in a clinical trial or use of an investigational drug within 30 days prior to admission to this study
16. Unwilling to discontinue use of an insulin pump for the duration of the study.
17. Women who are pregnant, nursing, or planning to become pregnant during the course of the study.
18. Patients on NPH as their basal insulin.
19. Positive history of hepatitis A (within 12 months of Screening), or a positive history of hepatitis B, hepatitis C, or HIV at Screening.
20. History of drug addiction and/or alcohol abuse within 12 months of Screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2016-06; Primary Completion 2018-04-28 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 26 weeks
  Change in HbA1c from Week 0 to Week 13, from Week 0 to Week 26, and from Week 13 to Week 26

SECONDARY OUTCOMES:
Change in fasting blood glucose glucose levels | 26 weeks
  Difference in fasting blood glucose levels Mean Mixed Tolerance Test AUC,
Hypoglycemia occurrences by category: Severe, Documented Symptomatic, and Asymptomatic Hypoglycemia | 26 weeks
  Comparison of frequency and severity of hypoglycemia
Number of Patients with Adverse Events | 26 weeks
  • To demonstrate the safety of HDV insulin lispro over 26 weeks of administration.
Change in total insulin usage | 26 weeks
  • Comparison of basal and bolus insulin doses as a mean of 3 days of use at Week 0 and at 13 and 26 weeks, and comparison of total bolus insulin dosing at end of run-in phase to the end of the 13 week treatment period, and from the 13 week treatment period to the 26 week treatment period.
Change in Body Weight | 26 weeks
  Comparison of change in body weight (in Kilograms) from baseline through week 26.
Mean Mixed Meal Tolerance Test | 13 and 26 weeks
  Comparison of mean mixed meal tolerance test (MMTT) (AUC0-120) from Week 0 (baseline) to Week 13, from Week 0 (baseline) to Week 26, and from Week 13 to Week 26

CONTACTS AND LOCATIONS:
Overall Officials: David Klonoff, MD, Principal Investigator — Mills-Peninsula Health Services
Locations (21):
- United States (21):
  - Hope & Wellness Clinical Trials, Inc., Corona, California
  - National Research Institute, Los Angeles, California
  - California Medical Research Associates Inc., Northridge, California
  - Bay Area Clinical Research, San Carlos, California
  - Mills-Peninsula Health Services, San Mateo, California
  - Orange County Research Center, Tustin, California
  - Creekside Endocrine Associates, PC, Denver, Colorado
  - Advanced Pharma CR, LLC, Miami, Florida
  - Ormond Medical Arts Pharmaceutical Research Center, Ormond Beach, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Rocky Mountain Diabetes & Osteoporosis Center, PA, Idaho Falls, Idaho
  - Associates in Endocrinology, Elgin, Illinois
  - University of Massachusetts Memorial Hospital, Worcester, Massachusetts
  - Desert Endocrinology Clinical Research Center, Henderson, Nevada
  - SUNY Upstate Medical University, Syracuse, New York
  - LION Research, Norman, Oklahoma
  - Endocrine and Psychiatry Center, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Rainier Clinical Research Center, Inc., Renton, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klonoff D, Bode B, Cohen N, Penn M, Geho WB, Muchmore DB. Divergent Hypoglycemic Effects of Hepatic-Directed Prandial Insulin: A 6-Month Phase 2b Study in Type 1 Diabetes. Diabetes Care. 2019 Nov;42(11):2154-2157. doi: 10.2337/dc19-0152. Epub 2019 Sep 24. PMID 31551249